CLINICAL TRIAL: NCT03027700
Title: Comparison of Non-invasive Methods to Detect and Quantify Liver Fibrosis
Brief Title: Methods to Detect Liver Fibrosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate recruitment
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: CIN001- Liver Fibrosis
Record Dates: First submitted 2017-01-19; First posted 2017-01-23 (Estimated); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Liver Fibroses; Hepatic Steatosis
MeSH Terms: conditions — Liver Cirrhosis; Fatty Liver

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Health/Normal Controls (Active Comparator): Health/normal control subjects will undergo MRI using several different imaging sequences (MR Elastography, T1 mapping, T2 mapping, T1 rho, and magnetization transfer) designed to detect and quantify hepatic fibrosis.
  Interventions: Device: MRI
- F1/F2 fibrosis (Active Comparator): Type 1 and 2 liver fibrosis subjects will undergo MRI using several different imaging sequences (MR Elastography, T1 mapping, T2 mapping, T1 rho, and magnetization transfer) designed to detect and quantify hepatic fibrosis.
  Interventions: Device: MRI
- F3/F4 fibrosis (Active Comparator): Type 2 and 3 liver fibrosis subjects will undergo MRI using several different imaging sequences (MR Elastography, T1 mapping, T2 mapping, T1 rho, and magnetization transfer) designed to detect and quantify hepatic fibrosis.
  Interventions: Device: MRI
- Hepatic steatosis with fibrosis (Active Comparator): Hepatic steatosis with liver fibrosis subjects will undergo MRI using several different imaging sequences (MR Elastography, T1 mapping, T2 mapping, T1 rho, and magnetization transfer) designed to detect and quantify hepatic fibrosis.
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — MRI scan performed on 1.5T Philips Ingenia MRI scanner.

SUMMARY:
The goal of this study is to learn more about liver fibrosis and methods to detect it. We will evaluate and compare multiple MRI based measures of liver fibrosis in subjects with and without liver disease.

DETAILED DESCRIPTION:
While liver biopsy is still considered the gold standard for diagnosing and assessing the presence and degree of liver fibrosis and inflammation, it has disadvantages including the potential for sampling error and risk of complications, including life-threatening bleeding. New imaging modalities such as MR Elastography, T1 mapping, T2 mapping, T1 rho, and magnetization transfer allow rapid, non-invasive evaluation of liver parenchymal characteristics and may be able to detect and quantify parenchymal fibrosis alleviating the need for biopsy. To date, the quantitative performance of these different techniques has not been extensively studied. This study is a single-center trial of non-invasive MR imaging techniques aimed at detecting and measuring liver fibrosis. Once optimized, these technologies may later be deployed in hypothesis driven research studies and/or routine clinical exams in the pediatric population here at CCHMC and/or as part of a multi-center study with specific IRB approval for that project.

To assess the relative performance of each technique, correlation across techniques, and reproducibility across the range of fibrosis, 32 subjects will be enrolled in this preliminary study sub-divided into 4 groups (Group 1: Healthy/ Normal controls; Group 2: F1/F2 fibrosis as determined by prior biopsy (low grade fibrosis group); Group 3: F3/F4 fibrosis as determined by prior biopsy (high grade fibrosis group), Group 4: Hepatic steatosis with fibrosis (NAFLD group)). 8 healthy subjects without known or suspected liver disease will be enrolled as normal controls. 8 subjects each with known fibrosis based on liver biopsy within the last 6 months will be enrolled in Group 2 and Group 3 (total = 16). 8 subjects with known hepatic steatosis and liver fibrosis based on liver biopsy within the last 6 months will be enrolled in Group 4.

ELIGIBILITY:
Inclusion Criteria

Group 1:

1. Healthy subjects with no known or suspected liver disease
2. Age 8 - 21 years

Groups 2 and 3:

1. Biopsy confirmed liver fibrosis (F1/F2 Group 2, F3/F4 Group 3)
2. Age 8 - 21 years

Group 4:

1. Biopsy confirmed hepatic steatosis AND biopsy confirmed liver fibrosis (any stage)
2. Age 8 - 21 years

Exclusion Criteria

All subjects:

1. Subjects <8 years of age and >21 years of age.
2. BMI > 35 kg/m2
3. Subjects deemed to possibly require sedation to undergo MR imaging
4. Inability to lie still for 90 minutes
5. Routine exclusions to MRI - e.g., implanted hardware
6. Pregnancy (verbal pregnancy screens - per standard practice in Radiology - will be administered to all female participants of child-bearing age at the time of enrollment and again immediately prior to imaging)
7. Prior history of liver transplantation

Group 1

1. ALT ≥30 U/L
2. Clinical history or lab/biopsy results suggestive of the presence of liver disease including: steatosis, fibrosis, inflammation, tumor, etc.

Group 2 and 3

1. Diagnosis of non-alcoholic fatty liver disease or non-alcoholic steatohepatitis
2. Biopsy >6 months prior to research MRI examination
3. Initiation of any medications (e.g. steroids, immunosuppressants, antivirals) or procedures (e.g. Kasai portoenterostomy) to treat the liver disease during the time between liver biopsy and study visit

Group 4

1. Biopsy >6 months prior to research MRI examination
2. Hepatic fat fraction >5%
3. Substantial weight loss (>10% of weight at time of biopsy) during the time between biopsy and study visit
4. Initiation of any medications to treat NAFLD (e.g. vitamin E) during the time between biopsy and study visit

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2017-01-26 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
MR imaging vs. histologic scoring in hepatic fibrosis | 2 years
  Correlate the results from the different imaging sequences designed to detect and quantify hepatic fibrosis

SECONDARY OUTCOMES:
MRI reproducibility | 2 years
  evaluate the reproducibility of each of the tested MRI-based liver fibrosis quantification sequences

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sporea I, Bota S, Jurchis A, Sirli R, Gradinaru-Tascau O, Popescu A, Ratiu I, Szilaski M. Acoustic radiation force impulse and supersonic shear imaging versus transient elastography for liver fibrosis assessment. Ultrasound Med Biol. 2013 Nov;39(11):1933-41. doi: 10.1016/j.ultrasmedbio.2013.05.003. Epub 2013 Aug 9. PMID 23932281
- [Background] Xanthakos SA, Podberesky DJ, Serai SD, Miles L, King EC, Balistreri WF, Kohli R. Use of magnetic resonance elastography to assess hepatic fibrosis in children with chronic liver disease. J Pediatr. 2014 Jan;164(1):186-8. doi: 10.1016/j.jpeds.2013.07.050. Epub 2013 Sep 21. PMID 24064151